CLINICAL TRIAL: NCT05841849
Title: Efficacy and Safety of Intravenous Versus Oral 5-HT3 Antagonists Combined With NK-1 Receptor Antagonists for the Prevention of Breast Cancer Chemotherapy-induced Nausea and Vomiting: a Single-center, Randomized Controlled Clinical Trial
Brief Title: Efficacy and Safety of Intravenous Versus Oral 5-HT3 Antagonists Combined With NK-1 Receptor Antagonists for the Prevention of CINV in Breast Cancer
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2023-0277
Record Dates: First submitted 2023-04-23; First posted 2023-05-03 (Actual); Last update posted 2023-05-03 (Actual); Status verified 2023-04

CONDITIONS: Breast Cancer; Chemotherapy-induced Nausea and Vomiting
Keywords: breast cancer; CINV; chemotherapy; oral versus intravenous
MeSH Terms: conditions — Breast Neoplasms; Vomiting | interventions — Aprepitant; Palonosetron; fosaprepitant

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- oral group (Experimental): patients receive oral palonosetron and aprepitant
  Interventions: Drug: Aprepitant; Drug: Palonosetron
- intravenous group (Active Comparator): patients receive intravenous palonosetron and fosaprepitant
  Interventions: Drug: Palonosetron; Drug: Fosaprepitant

INTERVENTIONS:
Drug: Aprepitant — oral aprepitant capsules 125mg for D1 before chemotherapy, 80mg for D2 and D3
  Arms: oral group
Drug: Palonosetron — oral palonosetron 0.5mg for D1 before chemotherapy; intravenous palonosetron 0.25mg for D1 before chemotherapy;
Drug: Fosaprepitant — intravenous fosaprepitant 150mg for D1 before chemotherapy
  Arms: intravenous group

SUMMARY:
Chemotherapy is one of the most common treatments for breast cancer, but the adverse effects can be severe enough to delay or make chemotherapy intolerable, thus affecting the efficacy of the disease. Women and younger patients are more likely to experience chemotherapy-induced nausea and vomiting (CINV) . Therefore, antiemetic drugs is a key way to reduce chemotherapy side effects, which ensures compliance, and maintain quality of life. CINV is usually induced by two pathways. The central pathway is mediated by neurokinin-1 (NK-1) receptors, where chemotherapeutic agents stimulate the secretion of substance-P (SP) from the vomiting center located in the medulla oblongata and nucleus accumbens, which binds to NK-1 receptors and induces vomiting. The peripheral pathway is mediated by 5-hydroxytryptamine 3 (5-HT3) receptors, and chemotherapy stimulates intestinal chromophores in the gastrointestinal mucosa to secrete 5-HT3, which binds to its receptors to induce vomiting.

Most guidelines currently recommend the combination of 5-HT3 receptor antagonists, NK-1 receptor antagonists, and dexamethasone for high-emetogenic-risk chemotherapy regimens. Usually 5-HT3 receptor antagonists include granisetron, ondansetron, and palonosetron. Palonosetron is a second-generation 5-HT3 receptor antagonist with stronger affinity and higher efficacy than other antagonists. The commonly used NK-1 receptor antagonists are aprepitant and fosaprepitant. Fosaprepitant is an aprepitant prodrug that can be rapidly converted to aprepitant in the body, blocking the binding of substance P to NK-1 receptors for antiemetic purposes. Clinical trial has confirmed that the overall complete response (CR) rate of palonosetron 0.75 mg combined with fosaprepitant and dexamethasone was 54.9%, with 75.9% CR in the acute phase (0-24 h after chemotherapy) and 62.3% in the delayed phase (24-72 h after chemotherapy). Another clinical trial showed an acute phase CR of 89.8% and a delayed phase CR of 90.4% for oral aprepitant combined with intravenous palonosetron 0.75 mg and dexamethasone. The data suggests that both oral and intravenous administration are effective in preventing CINV, but there are no clinical trial results for oral versus intravenous administration. Oral administration is painless, has fewer side effects, and is a safer mode of administration, but bioavailability is different and drug absorption is affected by a variety of factors; whereas intravenous injection has rapid onset of action, but there are risks of injection reactions, phlebitis, and infection. Therefore, we hope to conduct a non-inferiority study on the efficacy of oral and intravenous 5-HT3 receptor antagonists combined with NK-1 receptor antagonists through this trial, which can provide more options for patients by combining the cost and administration methods.

ELIGIBILITY:
Inclusion Criteria:

* Female, age 18-70 years.
* Confirmed pathology suggested primary invasive breast adenocarcinoma; Presence of adjuvant chemotherapy or neoadjuvant chemotherapy indications according to clinical guidelines.
* No other malignant tumor or other chemotherapy
* No prior treatment for present breast cancer onset
* ECOG physical status score 0 to 1
* Hematological examination before treatment should meet: white blood cell count (WBC) ≥ 4.0×10^9/L, neutrophil count (ANC) ≥ 1.5×10^9/L, platelet count (PLT) ≥ 100×10^9/L; hemoglobin (Hb) ≥ 90g/L; AST (sGOT), ALT (sGPT) ≤ 1.5 times the normal value upper limit, creatinine ≤ 1.5 times the upper limit of normal value, total bilirubin ≤ 1.5 times the upper limit of normal value.
* No serious impairment of heart, liver, kidney and other important organ functions.

Exclusion Criteria:

* Unwilling or unable to use an acceptable method of contraception for up to and including 8 weeks after the final dose of the test drug.
* Women during pregnancy and breastfeeding after pregnancy.
* Women with proven distant metastases of breast cancer.
* Patients with proven sensory or motor nerve disease.
* Definite cardiovascular disease, severe co-morbidity or active infection, including known HIV infection.
* Patients who need long-term anticoagulant drugs for cardiovascular or thrombotic diseases.
* History of other tumors.
* Allergic to the study drug or its excipients, etc.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1028 (Estimated)
Dates: Start 2023-07 (Estimated); Primary Completion 2028-07 (Estimated); Study Completion 2029-07 (Estimated)

PRIMARY OUTCOMES:
complete response | 0-72 hour after chemotherapy
  No vomiting or additional antiemetic medication throughout the post-chemotherapy period (0-72 hours)

SECONDARY OUTCOMES:
delayed phase complete response | 24-72 hour after chemotherapy
  Delayed phase (24-72 hours after chemotherapy) without vomiting or additional antiemetic medication use
acute phase complete response | 0-24 hour after chemotherapy
  Acute phase (0-24 hours after chemotherapy) without vomiting or additional antiemetic medication use

CONTACTS AND LOCATIONS:
Locations (1):
- the Second Affiliated Hospital of Zhejiang Univercity School of Medicine, Hanzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Navari RM, Aapro M. Antiemetic Prophylaxis for Chemotherapy-Induced Nausea and Vomiting. N Engl J Med. 2016 Apr 7;374(14):1356-67. doi: 10.1056/NEJMra1515442. No abstract available. PMID 27050207
- [Background] Gupta K, Walton R, Kataria SP. Chemotherapy-Induced Nausea and Vomiting: Pathogenesis, Recommendations, and New Trends. Cancer Treat Res Commun. 2021;26:100278. doi: 10.1016/j.ctarc.2020.100278. Epub 2020 Dec 11. PMID 33360668
- [Background] Hesketh PJ, Kris MG, Basch E, Bohlke K, Barbour SY, Clark-Snow RA, Danso MA, Dennis K, Dupuis LL, Dusetzina SB, Eng C, Feyer PC, Jordan K, Noonan K, Sparacio D, Lyman GH. Antiemetics: ASCO Guideline Update. J Clin Oncol. 2020 Aug 20;38(24):2782-2797. doi: 10.1200/JCO.20.01296. Epub 2020 Jul 13. PMID 32658626
- [Background] Navari RM. Palonosetron for the treatment of chemotherapy-induced nausea and vomiting. Expert Opin Pharmacother. 2014 Dec;15(17):2599-608. doi: 10.1517/14656566.2014.972366. Epub 2014 Oct 17. PMID 25323946
- [Background] Garnock-Jones KP. Fosaprepitant Dimeglumine: A Review in the Prevention of Nausea and Vomiting Associated with Chemotherapy. Drugs. 2016 Sep;76(14):1365-72. doi: 10.1007/s40265-016-0627-7. PMID 27510503
- [Background] Matsumoto K, Takahashi M, Sato K, Osaki A, Takano T, Naito Y, Matsuura K, Aogi K, Fujiwara K, Tamura K, Baba M, Tokunaga S, Hirano G, Imoto S, Miyazaki C, Yanagihara K, Imamura CK, Chiba Y, Saeki T. A double-blind, randomized, multicenter phase 3 study of palonosetron vs granisetron combined with dexamethasone and fosaprepitant to prevent chemotherapy-induced nausea and vomiting in patients with breast cancer receiving anthracycline and cyclophosphamide. Cancer Med. 2020 May;9(10):3319-3327. doi: 10.1002/cam4.2979. Epub 2020 Mar 13. PMID 32168551
- [Background] Nakayama Y, Ito Y, Tanabe M, Takahashi S, Hatake K. A combination of aprepitant, palonosetron, and dexamethasone prevents emesis associated with anthracycline-containing regimens for patients with breast cancer. A retrospective study. Breast Cancer. 2015 Mar;22(2):177-84. doi: 10.1007/s12282-013-0472-4. Epub 2013 May 8. PMID 23653153